CLINICAL TRIAL: NCT03015025
Title: Creation and Validation of a Pharmacogenetic Dosage Algorithm for Acenocoumarol in Patients With Venous Thromboembolic Disease, Atrial Fibrillation and/or Mechanical Valvular Heart Prosthesis
Brief Title: Pharmacogenetic Dosage Algorithm for Acenocoumarol
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: FC/HULP_005/2011
Record Dates: First submitted 2017-01-02; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2011-09

CONDITIONS: Atrial Fibrillation; Venous Thromboses; Cardiac Valve Disease
Keywords: Acenocoumarol; Cytochrome P450; Pharmacogenetics; Algorithm; CYP2C9; VKORC1; CYP4F2; P450 oxidoreductase (POR)
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Heart Valve Diseases; Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, Type 2 | interventions — Acenocoumarol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients' consent was requested for the preservation of their DNA sample, in case of new genes related to the pharmacokinetics or pharmacodynamics of acenocoumarol are discovered in the future.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stable treatment with acenocoumarol: Patients in stable anticoagulant treatment with acenocoumarol for auricular fibrillation, venous thromboembolic disease and/or cardiac valve replacement.
  Interventions: Genetic: Acenocoumarol

INTERVENTIONS:
Genetic: Acenocoumarol — A blood sample was collected for CYP2C9, VKORC1, CYP4F2, APOE and 2 variants of POR genotypes.

SUMMARY:
The use of coumarins has been a challenge for doctors because of its narrow therapeutic range and they show great inter and intra-individual variability in the dose necessary to achieve an international normalized ratio (INR) within the therapeutic range. Among the factors influencing the interindividual variability in the dose required include age, weight, Vitamin K in the diet, comorbidity as well as drug interactions and in recent years has also seen the importance of pharmacogenetic factors.

DETAILED DESCRIPTION:
Demographic and clinical factors contribute approximately 20% to the total variability of dose requirements. In recent years it has highlighted the close relationship between the dose requirements of coumarin drugs and certain polymorphisms of genes involved in pharmacokinetics and pharmacodynamics of these drugs. The use of dosing algorithms that include pharmacogenetic information may help in the dose selection, improving efficacy and reducing adverse events. Studies have shown the relationship between genotype variants of CYP2C9 and VKORC1, CYP4F2 and apolipoprotein E (ApoE), which together with the demographic and clinical variants can explain between 50-60% of the variability in the response to these drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Auricular fibrillation, venous thromboembolic disease and cardiac valve replacement receiving acenocoumarol.
* Patients with stable dose of acenocoumarol (weekly dose variation of <20% in the last 3 months).
* Patients with an international normalised ratio within the range of 2 to 3 (in Auricular Fibrillation and venous thromboembolic disease) or 2.5 to 3.5 (in cardiac valve replacement) for at least the 3 previous consecutive months.

Exclusion Criteria:

* Patients with renal failure (calculated creatinine clearance ≤30 ml/min), hepatic disease (stage C of Child Plough Stage), thyroid dysfunction and/or cancer.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving stable anticoagulant treatment with acenocoumarol for auricular fibrillation, venous thromboembolic disease and/or cardiac valve replacement in Hospital La Paz and Barrio del Pilar primary care center.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Creation of a pharmacogenetic algorithm of dosage for acenocoumarol | Up to 5 years

SECONDARY OUTCOMES:
Validation of the pharmacogenetic algorithm. | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carcas, MD, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No